CLINICAL TRIAL: NCT07362966
Title: Effect of Colchicine on Progression of Coronary Atherosclerosis in Patients With TET2-CHIP Variant: a Pilot Clinical Trial (COLCHIP-Pilot)
Brief Title: Effect of Colchicine on Progression of Coronary Atherosclerosis in Patients With TET2-CHIP Variant
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, MD, PhD, Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COLCHIP-Pilot
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Colchicine; Coronary Atherosclerosis Management; Clonal Hematopoiesis of Indeterminate Potential
MeSH Terms: interventions — Colchicine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Colchicine with SoC therapy (TET2-CHIP group) (Experimental): Participants with TET2-CHIP will receive colchicine 0.5 mg orally once daily plus standard of care (SoC) therapy for 12 months.
  Interventions: Drug: Colchicine 0.5 mg orally once daily for 12 months.; Other: SoC therapy
- SoC therapy alone (TET2-CHIP group) (No Intervention): Participants with TET2-CHIP will receive SoC therapy alone (no colchicine) for 12 months.
- Colchicine with SoC therapy (non-CHIP group) (Experimental): Participants without CHIP-associated variants will receive colchicine 0.5 mg orally once daily plus standard of care (SoC) therapy for 12 months.
  Interventions: Drug: Colchicine 0.5 mg orally once daily for 12 months.; Other: SoC therapy
- SoC therapy alone (non-CHIP group) (No Intervention): Participants without CHIP-associated variants will receive SoC therapy alone (no colchicine) for 12 months.

INTERVENTIONS:
Drug: Colchicine 0.5 mg orally once daily for 12 months. — SoC therapy includes but is not limited to appropriate lipid lowering, anti-platelet therapy, anti-hypertensive and beta blockers as defined by local guidelines.
  Arms: Colchicine with SoC therapy (TET2-CHIP group); Colchicine with SoC therapy (non-CHIP group)
Other: SoC therapy — SoC therapy
  Arms: Colchicine with SoC therapy (TET2-CHIP group); Colchicine with SoC therapy (non-CHIP group)

SUMMARY:
This study aims to investigate whether TET2-associated clonal hematopoiesis of indeterminate potential (TET2-CHIP) can serve as a biomarker to guide precision use of colchicine in a population of clinically stable post-ACS patients receiving standard of care (SoC) therapy. Specifically, we will evaluate whether TET2-CHIP status predicts a differential response to colchicine. As a pilot study, it also aims to provide detailed data supporting design of further trial, such as sample size calculating, endpoint optimizing, etc.

DETAILED DESCRIPTION:
COLCHIP-Pilot is a single-center, prospective, randomized, open-label, assessor-blinded pilot trial. A total of 120 patients will be enrolled and stratified by CHIP variant status into a TET2-CHIP group or a non-CHIP group. TET2-CHIP group (N = 60): Participants will be randomized (1:1) to colchicine 0.5 mg once daily plus SoC therapy (n = 30) or SoC therapy alone (control; n = 30). Non-CHIP group (N = 60): Participants will be randomized (1:1) to colchicine 0.5 mg once daily plus SoC therapy (n = 30) or SoC therapy alone (control; n = 30). SoC therapy includes but is not limited to appropriate lipid lowering, anti-platelet therapy, anti-hypertensive and beta blockers as defined by local guidelines. Patients should also be instructed to follow heart healthy (low fat) diet and regular exercise program. The index qualifying ACS must have occurred at least 30 days and no more than 90 days prior to randomization.

Baseline assessment for all participants will include coronary CT angiography (CCTA) using photon-counting detector CT (PCD-CT), inflammatory biomarkers testing and CHIP variant sequencing. After randomization, participants will have visits at Month 0, 1, 3, 6, 9, and 12. Repeat CCTA for the assessment of coronary plaque will occur during the Month 12 visit. The primary endpoint is the percent change in total plaque volume in non-culprit coronary lesion from baseline to Month 12, measured by CCTA. Secondary endpoints include the percent change in other plaques (calcified plaque, noncalcified plaque, low attenuation plaque, and fibrotic plaque) volume of coronary artery plaque from baseline to Month 12; change in levels of inflammatory biomarkers (IL-6, IL-1β, IL-18, hs-CRP, and S100A12); change in the TET2-CHIP variant allele fraction; and major adverse cardiovascular events (MACE), defined as a composite of all-cause death, nonfatal myocardial infarction, nonfatal stroke, and ischemia-driven revascularization. Participants will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-85 years;
2. Patients with recent hospitalization for documented ACS (the index event occurring 30-90 days before randomization) and meeting all of the following:

   1. During the index hospitalization, patients underwent either PCI or diagnostic coronary angiography alone,
   2. At least one non-culprit coronary lesion with 30%-70% diameter stenosis by visual estimation on coronary angiography,
   3. Clinically stable throughout the screening period,
   4. Receiving standard of care therapy for ACS in accordance with national guidelines,
   5. Peripheral blood DNA available for targeted sequencing, with results demonstrating either TET2-CHIP or no CHIP-associated variants;
3. Written informed consent.

Exclusion Criteria:

1. Prior PCI or coronary artery bypass grafting (CABG) before documented ACS;
2. Other clinically significant cardiovascular diseases, including moderate-to-severe valvular heart disease (moderate or severe), heart failure (NYHA class III-IV), or atrial fibrillation;
3. Non-culprit coronary anatomy (e.g., marked tortuosity, bifurcation lesions, or small vessels <1.5 mm in diameter) deemed to preclude plaque assessment by CCTA;
4. Planned PCI or CABG;
5. Abnormal liver function (ALT >3 times the upper limit of normal range) at randomization;
6. Abnormal renal function (serum creatinine >1.5 times the upper limit of normal range or estimated eGFR <45 mL/min/1.73 m²) at randomization;
7. Hematologic abnormalities: anemia (hemoglobin <100g/L), thrombocytopenia (platelet count <100×109/L) or leukopenia (white blood cell <3×109/L) at randomization;
8. Inflammatory bowel disease (Crohn's or ulcerative colitis) or active diarrhea;
9. Symptomatic peripheral neuropathy, pre-existing progressive neuromuscular disease or creatine kinase (CK) level > 3 times the upper limit of normal range as measured within the past 30 days and determined to be non-transient through repeat testing;
10. Pregnancy, breastfeeding, or women of childbearing potential who are not using an effective method of contraception;
11. Any contraindication, known allergy or intolerance to colchicine;
12. Colchicine use within 30 days prior to randomization, or planned colchicine therapy for other indications;
13. Current or planned use of any of cyclosporine, verapamil, HIV protease inhibitors, azole antifungals, or macrolide antibiotics;
14. Existing or planned treatment with other anti-inflammatory or immunosuppressive drugs;
15. History of malignancy (hematologic or solid-tumor);
16. History of transplantation (hematopoietic stem cell or solid-organ);
17. Significant radiation exposure (≥40 mSv) within the past 12 months;
18. Known hypersensitivity to iodinated contrast media or uncontrolled active hyperthyroidism;
19. Current enrollment in another clinical trial;
20. A predicted life expectancy < 1 year;
21. Any other circumstances in which the investigator judges that the patient is not suitable to participate in the clinical trial.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-02-24 (Estimated); Primary Completion 2027-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Percent change in total plaque volume of coronary artery plaque | Up to 12 months
  Percent change in total plaque volume of coronary artery plaque measured by CCTA

SECONDARY OUTCOMES:
Percent change in other plaques (calcified plaque, noncalcified plaque, low attenuation plaque, and fibrotic plaque) volume of coronary artery plaque | Up to 12 months
  Percent change in other plaques (calcified plaque, noncalcified plaque, low attenuation plaque, and fibrotic plaque) volume of coronary artery plaque measured by CCTA.
Change in levels of inflammatory biomarkers | Up to 12 months
  Change in levels of circulating IL-6, IL-1β, IL-18, hs-CRP, and S100A12.
Change in TET2-CHIP variant allele fraction at 6 months | Up to 6 months
  Change in TET2-CHIP variant allele fraction measured by next generation sequencing.
Change in TET2-CHIP variant allele fraction at 12 months | Up to 12months
  Change in TET2-CHIP variant allele fraction measured by next generation sequencing.
Major adverse cardiovascular events (MACE) | Up to 12 months
  A composite of all-cause death, nonfatal myocardial infarction, nonfatal stroke, and ischemia-driven revascularization.

CONTACTS AND LOCATIONS:
Overall Officials: Yaling Han, MD, PhD, Study Chair — The General Hospital of Northern Theater Command
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No